CLINICAL TRIAL: NCT06467305
Title: Sensorimotor Basis of Speech Motor Learning and Retention
Brief Title: Speech Motor Learning and Retention (Aim 1)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000037622_a; 1R01DC022097-01A1 (NIH)
Record Dates: First submitted 2024-06-13; First posted 2024-06-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Speech
Keywords: Speech Motor Learning; Retention
MeSH Terms: conditions — Speech | interventions — Acclimatization

STUDY DESIGN:
Intervention Model Description: Healthy right-handed adults with normal hearing will be recruited in equal number from both sexes. All participants will be fluent English speakers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Altered auditory feedback + cTBS to auditory cortex (Experimental): Participants will perform learning tasks while receiving altered auditory feedback.This procedure will be repeated on day 2. cTBS will be applied to the left hemisphere auditory cortex following learning. Participants then leave the laboratory and return 24 hours later to assess retention of learning.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation
- Altered auditory feedback + cTBS to somatosensory cortex (Experimental): Participants will perform learning tasks while receiving altered auditory feedback.This procedure will be repeated on day 2. cTBS will be applied to the left hemisphere somatosensory cortex following learning. Participants then leave the laboratory and return 24 hours later to assess retention of learning.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation
- Altered auditory feedback + cTBS to motor cortex (Experimental): Participants will perform learning tasks while receiving altered auditory feedback.This procedure will be repeated on day 2. cTBS will be applied to the left hemisphere motor cortex following learning. Participants then leave the laboratory and return 24 hours later to assess retention of learning.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation
- Altered auditory feedback + cTBS to motor cortex control zone (Experimental): Participants in a control condition will undergo the same procedures using cTBS to a motor cortex control zone in the right hemisphere (associated with the hand muscle first dorsal interosseous). cTBS will be applied following learning and subjects will return 24 hours later to test for retention. This control condition is included as a test for non-specific effects of cTBS stimulation.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation
- Unaltered auditory feedback + cTBS to auditory cortex (Experimental): Participants will perform learning tasks while receiving unaltered auditory feedback.This procedure will be repeated on day 2. cTBS will be applied to the left hemisphere auditory cortex following learning. Participants then leave the laboratory and return 24 hours later to assess retention of learning. If the effects of cTBS are specific to learning, no effect should be observed in these control conditions.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation
- Unaltered auditory feedback + cTBS to somatosensory cortex (Experimental): Participants will perform learning tasks while receiving unaltered auditory feedback.This procedure will be repeated on day 2. cTBS will be applied to the left hemisphere somatosensory cortex following learning. Participants then leave the laboratory and return 24 hours later to assess retention of learning. If the effects of cTBS are specific to learning, no effect should be observed in these control conditions.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation
- Unaltered auditory feedback + cTBS to motor cortex (Experimental): Participants will perform learning tasks while receiving unaltered auditory feedback.This procedure will be repeated on day 2. cTBS will be applied to the left hemisphere motor cortex following learning. Participants then leave the laboratory and return 24 hours later to assess retention of learning. If the effects of cTBS are specific to learning, no effect should be observed in these control conditions.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation
- Unaltered auditory feedback + cTBS to motor cortex control zone (Experimental): Participants in a control condition will undergo the same procedures using cTBS to a motor cortex control zone in the right hemisphere (associated with the hand muscle first dorsal interosseous). cTBS will be applied following learning and subjects will return 24 hours later to test for retention. This control condition is included as a test for non-specific effects of cTBS stimulation. If the effects of cTBS are specific to learning, no effect should be observed in these control conditions.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation

INTERVENTIONS:
Device: continuous theta-burst stimulation (cTBS) — Non-invasive brain stimulation, evoked potentials and fMRI will be used to identify brain regions involved in speech motor learning and retention.
Behavioral: Adaptation — Auditory adaptation in speech

SUMMARY:
The overall goal of this research is to test a new model of speech motor learning, whose central hypothesis is that learning and retention are associated with plasticity not only in motor areas of the brain but in auditory and somatosensory regions as well. The strategy for the proposed research is to identify individual brain areas that contribute causally to retention by disrupting their activity with transcranial magnetic stimulation (TMS). Investigators will also use functional magnetic resonance imaging (fMRI) which will enable identification of circuit-level activity which predicts either learning or retention of new movements, and hence test the specific contributions of candidate sensory and motor zones. In other studies, investigators will record sensory and motor evoked potentials over the course of learning to determine the temporal order in which individual sensory and cortical motor regions contribute. The goal here is to identify brain areas in which learning-related plasticity occurs first and which among these areas predict subsequent learning.

DETAILED DESCRIPTION:
The focus of this registration is Aim 1. The work in Specific Aim 1 involves tests of speech motor memory retention following disruption of left hemisphere brain activity in either auditory, somatosensory or motor cortex or to a control site (hand area motor cortex right hemisphere). Continuous theta-burst stimulation (cTBS) is delivered following adaptation to altered auditory feedback to assess its effects on the retention of new learning. In the adaptation task, participants read Harvard Sentences aloud, which are presented on a computer monitor. Vocal output is altered in real-time and played back to participants through headphones. Tests of retention are conducted 24 hours later.

The Speech Motor Learning and Retention Master Protocol has uniqueID 2000037622.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speakers
* Right-handed
* Normal hearing
* No speech disorder or reading disability

Exclusion Criteria:

* Cardiac pacemaker
* Aneurysm clip
* Heart or Vascular clip
* Prosthetic valve
* Metal implants
* Metal in brain, skull, or spinal cord
* Implanted neurostimulator
* Medication infusion device
* Cochlear implant or tinnitus (ringing in ears)
* Personal and/or family history of epilepsy or other neurological disorders or history of head concussion
* Psychoactive medications
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Speech motor learning | Performance as measured at the end of learning (30 minute session)
  Audapter software will be used to alter the first and second formant frequencies of the spoken words and this is played back to subjects through headphones. Subjects will be tested both with unaltered feedback and with abruptly introduced frequency shifts.The change in the first (F1) and second format frequency (F2) values will be assessed using Praat.
Retention of learning | 24 hours after learning (re-test lasts 30 minutes)
  The retention of adaptation to altered auditory feedback (and relearning) will be quantified in terms of F1 and F2 frequency shifts (relative to pre-training baseline). Larger values indicate more complete relearning or retention.

CONTACTS AND LOCATIONS:
Overall Officials: David Ostry, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No